CLINICAL TRIAL: NCT03370939
Title: Endovascular Treatment Key Technique and Emergency Work Flow Improvement of Acute Ischemic stroke-a Prospective Multicenter Registry Study
Brief Title: Endovascular Treatment Key Technique and Emergency Work Flow Improvement of Acute Ischemic Stroke
Acronym: ANGEL-ACT
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Director, Department of interventional neurology, Beijing Tiantan Hospital
Other Study IDs: 2016YFC1301501-1
Record Dates: First submitted 2017-10-18; First posted 2017-12-13 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Intracranial Artery Occlusion With Infarction (Disorder)
Keywords: ischemic stroke; endovascular treatment; registry
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endovascular thrombectomy (EVT) is effective and safe for acute ischemic stroke (AIS) caused by large vessel occlusion (LVO) in major clinical trials. Whether the benefit of EVT in randomized trials could be generalized to clinical practice, especially in developing countries, remains unknown. The prospective Chinese ANGEL-ACT Registry (Endovascular Treatment Key Technique and Emergency Work Flow Improvement of Acute Ischemic Stroke) was established to evaluate the utilization, and subsequent outcomes of EVT treated AIS patients. This study is a multi-center, prospective registry study initiated by researchers, funded by National Key R&D Program of China. A total of 2,000 patients with acute ischemic stroke will undergo endovascular treatment. The hypothesis was that favorable outcomes from clinical trials could be achieved in clinical practice in China.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years old;
2. Diagnosis of acute ischemic stroke;
3. Imaging confirmed intracranial large artery occlusion (LVO): intracranial internal carotid artery (ICA T/L), middle cerebral artery (MCA M1/M2), anterior cerebral artery (ACA A1/A2), basilar artery (BA), vertebral artery (VA V4), and posterior cerebral artery (PCA P1);
4. Initiation of any type of endovascular treatment (EVT), including intra-arterial thrombolysis, mechanical thrombectomy, angioplasty, and stenting;
5. The patient or the patient's legal representative is able and willing to sign the informed consent.

Exclusion criteria

1. Isolated cervical ICA or VA occlusion;
2. No evidence of LVO on DSA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke caused by large vessel occlusion and receiving endovascular treatment.
Sampling Method: Non-Probability Sample
Enrollment: 2004 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Functional independence at 90 days (modified Rankin Scale of 0-2) | 90±7 days after enrollment
  The range of modified Rankin Scale was from 0 to 6. 0-No symptoms;1-No significant disability;2-Slight disability;3-Moderate disability;4-Moderately severe disability;5-Severe disability;6 -Dead.A higher score indicates worse a outcome.
Symptomatic intracranial hemorrhage (sICH) within 12-36 hours after the procedure | 12-36 hours after the procedure
  Heidelberg Bleeding Classification): new intracranial hemorrhage detected by brain imaging associated with ≥4 points total National Institutes of Health Stroke Scale (NIHSS), ≥2 points in one NIHSS category, leading to intubation/ hemicraniectomy/ EVD placement or other major medical/surgical intervention, or absence of alternative explanation for deterioration
Time from symptom onset to recanalization | The end of the procedure

SECONDARY OUTCOMES:
Recanalization rate at the end of the procedure | at the end of the procedure
  mTICI score 2b-3
Recanalization rate after the first attempt | At baseline, during the procedure, after the first attempt of endovascular treatment
  mTICI score 2b-3
Changes in NIHSS score immediately after the procedure | within 2 hours after the procedure
  difference between NIHSS score immediately after the procedure and baseline
Changes in NIHSS score 24 hours after the procedure | 24 hours after the procedure
  difference between NIHSS score 24 hours after the procedure and baseline
Changes in NIHSS score 7 days after the procedure or at discharge | 7 days after the procedure or discharge
  difference between NIHSS score 7 days after the procedure or discharge and baseline
EQ-5D 90 days after the procedure | 90±7 days after the procedure
  EQ-5D is a standardized instrument for measuring generic health status. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).A higher score indicates a better outcome.
Barthel index (BI) 90 days after the procedure | 90±7 days after the procedure
  The BI has a score of 0-100. A higher score indicates a better outcome.
Parenchymal hematoma (PH2) | 12-36 hours after the procedure
  PH2 is defined as hematoma in >30% of infarct area
Any intracranial hemorrhage on imaging | 12-36 hours after the procedure
All-cause mortality within 90 days | 90±7 days after the procedure
Time from onset to arrival | At baseline, after arrival at the hospital
Time from arrival to imaging | At baseline, after taking any brain imaging
Time from imaging to puncture | At baseline, during the procedure, after successful groin puncture
Time from puncture to recanalization | At baseline, during the procedure, after successful recanalization

CONTACTS AND LOCATIONS:
Overall Officials: Zhongrong Miao, PhD, Principal Investigator — Capital Medical University, Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Bu Z, Sun D, Zhang X, Ma N, Gao F, Mo D, Meng Q, Miao Z; ANGEL-ACT study group. The role of intravenous tirofiban in patients undergoing endovascular treatment for acute intracranial atherosclerotic occlusion. J Stroke Cerebrovasc Dis. 2025 Oct;34(10):108420. doi: 10.1016/j.jstrokecerebrovasdis.2025.108420. Epub 2025 Aug 11. PMID 40803585
- [Derived] Tong X, Jia B, Ma G, Zhang X, Fiehler J, Flottmann F, Bechstein M, Broocks G, Hanning U, Kniep HC, Thomalla G, Deb-Chatterji M, Schon G, Zhang Y, Gao F, Ma N, Mo D, Miao Z, Meyer L; as the ANGEL-ACT & GSR-ET study group. Relationship Between Thrombolysis-to-Puncture Time and Outcomes of Endovascular Thrombectomy in Acute Ischemic Stroke. Neurol Clin Pract. 2025 Aug;15(4):e200434. doi: 10.1212/CPJ.0000000000200434. Epub 2025 Jul 11. PMID 40656129
- [Derived] Bu Z, Sun D, Ma G, Jia B, Tong X, Huo X, Wang A, Ma N, Gao F, Mo D, Song L, Sun X, Deng Y, Li X, Wang B, Luo G, Su D, Miao Z. The impact of intraarterial, intravenous, and combined tirofiban on endovascular treatment for acute intracranial atherosclerotic occlusion. Front Neurol. 2024 Feb 13;15:1336098. doi: 10.3389/fneur.2024.1336098. eCollection 2024. PMID 38414555
- [Derived] Li L, Lv J, Han JJ, Gao Y, Yan ZX, Wu Q, Zhang XL, Gao F. Nomogram model of functional outcome for endovascular treatment in patients with acute basilar artery occlusion. Front Neurol. 2023 Oct 19;14:1277189. doi: 10.3389/fneur.2023.1277189. eCollection 2023. PMID 37928150
- [Derived] Deng Y, Yao Y, Tong X, Yin Y, Wang A, Zhang Y, Jia B, Huo X, Luo G, Ma N, Mo D, Song L, Sun X, Gao F, Chen D. Necessity and timing of angioplasty in acute large-vessel occlusion strokes due to intracranial atherosclerotic disease: A cohort analysis with data from the angel-ACT registry. Front Neurol. 2023 Mar 16;14:1087816. doi: 10.3389/fneur.2023.1087816. eCollection 2023. PMID 37006506
- [Derived] Sun D, Huo X, Raynald, Jia B, Tong X, Wang A, Ma N, Gao F, Mo D, Miao Z; ANGEL-ACT study group. First pass effect of mechanical thrombectomy for acute vertebrobasilar artery occlusion: data from the ANGEL-ACT registry. J Neurointerv Surg. 2023 Dec;15(12):1201-1206. doi: 10.1136/jnis-2023-020065. Epub 2023 Feb 1. PMID 36725361
- [Derived] Sun D, Raynald, Huo X, Jia B, Tong X, Ma G, Wang A, Ma N, Gao F, Mo D, Nguyen TN, Miao Z; ANGEL-ACT Study Group. Sex-Related Differences in Outcomes of Endovascular Treatment for Anterior Circulation Large Vessel Occlusion. Stroke. 2023 Feb;54(2):327-336. doi: 10.1161/STROKEAHA.122.041195. Epub 2023 Jan 23. PMID 36689588
- [Derived] Li K, Sun D, Tong X, Wang A, Zhang Y, Ma G, Huo X, Ma N, Gao F, Mo D, Sun X, Peng G, Zhang X, Jia B, Miao Z. Incidence, predictors, and impact on outcome of underlying intracranial atherosclerotic disease in acute vertebrobasilar artery occlusion undergoing endovascular therapy: Data from ANGEL-ACT registry. Int J Stroke. 2023 Aug;18(7):856-863. doi: 10.1177/17474930221150111. Epub 2023 Jan 14. PMID 36571164
- [Derived] Sun D, Huo X, Raynald, Wang A, Jia B, Tong X, Ma G, Mo D, Gao F, Ma N, Miao Z. Predictors of poor outcome after endovascular treatment for acute vertebrobasilar occlusion: data from ANGEL-ACT registry. Neuroradiology. 2023 Jan;65(1):177-184. doi: 10.1007/s00234-022-03065-x. Epub 2022 Oct 24. PMID 36274108
- [Derived] Tong X, Burgin WS, Ren Z, Jia B, Zhang X, Huo X, Luo G, Wang A, Zhang Y, Ma N, Gao F, Song L, Sun X, Liu L, Deng Y, Li X, Wang B, Ma G, Wang Y, Wang Y, Miao Z, Mo D; ANGEL-ACT Study Group. Association of Stroke Subtype With Hemorrhagic Transformation Mediated by Thrombectomy Pass: Data From the ANGEL-ACT Registry. Stroke. 2022 Jun;53(6):1984-1992. doi: 10.1161/STROKEAHA.121.037411. Epub 2022 Mar 31. PMID 35354298
- [Derived] Raynald, Sun D, Huo X, Jia B, Tong X, Ma G, Wang A, Mo D, Ma N, Gao F, Amin S, Ren Z, Miao Z; ANGEL-ACT study group. The Safety and Efficacy of Endovascular Treatment in Acute Ischemic Stroke Patients Caused by Large-Vessel Occlusion with Different Etiologies of Stroke: Data from ANGEL-ACT Registry. Neurotherapeutics. 2022 Mar;19(2):501-512. doi: 10.1007/s13311-022-01189-9. Epub 2022 Mar 3. PMID 35243592
- [Derived] Ma G, Sun X, Cheng H, Burgin WS, Luo W, Jia W, Liu Y, He W, Geng X, Zhu L, Chen X, Shi H, Xu H, Zhang L, Wang A, Mo D, Ma N, Gao F, Song L, Huo X, Deng Y, Liu L, Luo G, Jia B, Tong X, Liu L, Ren Z, Miao Z; EPOCH Study and ANGEL-ACT Study Groups. Combined Approach to Eptifibatide and Thrombectomy in Acute Ischemic Stroke Because of Large Vessel Occlusion: A Matched-Control Analysis. Stroke. 2022 May;53(5):1580-1588. doi: 10.1161/STROKEAHA.121.036754. Epub 2022 Feb 2. PMID 35105182
- [Derived] Sun D, Jia B, Tong X, Kan P, Huo X, Wang A, Raynald, Ma G, Ma N, Gao F, Mo D, Song L, Sun X, Liu L, Deng Y, Li X, Wang B, Luo G, Wang Y, Ren Z, Miao Z; ANGEL-ACT study group. Predictors of parenchymal hemorrhage after endovascular treatment in acute ischemic stroke: data from ANGEL-ACT Registry. J Neurointerv Surg. 2023 Jan;15(1):20-26. doi: 10.1136/neurintsurg-2021-018292. Epub 2022 Jan 12. PMID 35022299
- [Derived] Ding Y, Gao F, Ji Y, Zhai T, Tong X, Jia B, Wu J, Wu J, Zhang Y, Wei C, Wang W, Zhou J, Niu J, Miao Z, Liu Y. Workflow Intervals and Outcomes of Endovascular Treatment for Acute Large-Vessel Occlusion During On-Vs. Off-hours in China: The ANGEL-ACT Registry. Front Neurol. 2021 Dec 21;12:771803. doi: 10.3389/fneur.2021.771803. eCollection 2021. PMID 34992575
- [Derived] Huo X, Sun D, Raynald, Jia B, Tong X, Wang A, Ma N, Gao F, Mo D, Ma G, Amin S, Ren Z, Miao Z; ANGEL-ACT study group. Endovascular Treatment in Acute Ischemic Stroke with Large Vessel Occlusion According to Different Stroke Subtypes: Data from ANGEL-ACT Registry. Neurol Ther. 2022 Mar;11(1):151-165. doi: 10.1007/s40120-021-00301-z. Epub 2021 Nov 20. PMID 34800279
- [Derived] Sun D, Tong X, Huo X, Jia B, Raynald, Wang A, Ma G, Ma N, Gao F, Mo D, Song L, Sun X, Liu L, Deng Y, Li X, Wang B, Luo G, Wang Y, Miao Z; ANGEL-ACT study group. Unexplained early neurological deterioration after endovascular treatment for acute large vessel occlusion: incidence, predictors, and clinical impact: Data from ANGEL-ACT registry. J Neurointerv Surg. 2022 Sep;14(9):875-880. doi: 10.1136/neurintsurg-2021-017956. Epub 2021 Sep 30. PMID 34593600
- [Derived] Tong X, Li S, Liu W, Ren Z, Liu R, Jia B, Zhang X, Huo X, Luo G, Ma G, Wang A, Wang Y, Wang Y, Miao Z, Mo D; ANGEL-ACT study group. Endovascular treatment for acute ischemic stroke in patients with versus without atrial fibrillation: a matched-control study. BMC Neurol. 2021 Sep 29;21(1):377. doi: 10.1186/s12883-021-02386-3. PMID 34587913
- [Derived] Tong X, Wang Y, Bauer CT, Jia B, Zhang X, Huo X, Luo G, Wang A, Ma N, Gao F, Mo D, Song L, Sun X, Liu L, Deng Y, Li X, Wang B, Ma G, Wang Y, Ren Z, Miao Z. Current status of aspiration thrombectomy for acute stroke patients in China: data from ANGEL-ACT Registry. Ther Adv Neurol Disord. 2021 Apr 12;14:17562864211007715. doi: 10.1177/17562864211007715. eCollection 2021. PMID 33912244
- [Derived] Tong X, Wang Y, Fiehler J, Bauer CT, Jia B, Zhang X, Huo X, Luo G, Wang A, Pan Y, Ma N, Gao F, Mo D, Song L, Sun X, Liu L, Deng Y, Li X, Wang B, Ma G, Wang Y, Ren Z, Miao Z; ANGEL-ACT Study Group. Thrombectomy Versus Combined Thrombolysis and Thrombectomy in Patients With Acute Stroke: A Matched-Control Study. Stroke. 2021 May;52(5):1589-1600. doi: 10.1161/STROKEAHA.120.031599. Epub 2021 Mar 4. PMID 33657849
- [Derived] Jia B, Ren Z, Mokin M, Burgin WS, Bauer CT, Fiehler J, Mo D, Ma N, Gao F, Huo X, Luo G, Wang A, Pan Y, Song L, Sun X, Zhang X, Gui L, Song C, Peng Y, Wu J, Zhao S, Zhao J, Zhou Z, Li Y, Jing P, Yang L, Liu Y, Zhao Q, Liu Y, Peng X, Gao Q, Guo Z, Chen W, Li W, Cheng X, Xu Y, Zhang Y, Zhang G, Lu Y, Lu X, Wang D, Wang Y, Li H, Ling L, Peng G, Zhang J, Zhang K, Li S, Qi Z, Xu H, Tong X, Ma G, Liu R, Guo X, Deng Y, Leng X, Leung TW, Liebeskind DS, Wang Y, Wang Y, Miao Z; ANGEL-ACT Study Groupdagger. Current Status of Endovascular Treatment for Acute Large Vessel Occlusion in China: A Real-World Nationwide Registry. Stroke. 2021 Apr;52(4):1203-1212. doi: 10.1161/STROKEAHA.120.031869. Epub 2021 Feb 18. PMID 33596674